CLINICAL TRIAL: NCT04974684
Title: Direct Oral Anticoagulant Therapy With the HeartMate 3 LVAD: A Pilot Study
Brief Title: DOT HeartMate 3 Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Prof. Ivan Netuka, MD, Ph.D., Chairman of the Cardiovascular Surgery Department, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A-21-23
Record Dates: First submitted 2021-06-23; First posted 2021-07-23 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: LVAD (Left Ventricular Assist Device) Thrombosis
Keywords: HeartMate 3; LVAD (Left Ventricular Assist Device); NOAC
MeSH Terms: conditions — Thrombosis | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Interventional group (Experimental): This study group will contain 30 patients that will be stratified further by 1:1 randomization to 2 groups of 15 patients - one group will be given only apixaban 5mg twice a day, the second group will be given apixaban 5mg twice a day and aspirin 100mg per day.
  Interventions: Device: HeartMate 3; Drug: Apixaban
- Control group (No Intervention): This study group will contain 15 patients that will by treated following standard anticoagulation protocol (Warfarin INR 2-3 + aspirin 100mg/day).

INTERVENTIONS:
Device: HeartMate 3 — Patients implanted with HeartMate 3 will be randomized in 2:1 ratio in interventional and control group. Patients in interventional group will be switched to therapy with apixaban instead of warfarin.
  Arms: Interventional group
Drug: Apixaban — Patients implanted with HeartMate 3 will be randomized in 2:1 ratio in interventional and control group. Patients in interventional group will be switched to therapy with apixaban instead of warfarin.
  Arms: Interventional group

SUMMARY:
A prospective, single-center, randomized controlled trial of the feasibility and safety of apixaban in HeartMate 3 patients.

DETAILED DESCRIPTION:
HeartMate 3 (HM3) Left Ventricular Assist System (LVAS) is a centrifugal, fully magnetically levitated, continuous-flow pump designed to facilitate hemocompatibility by reducing shear stress on blood elements and to optimize pump washout by intrinsic pulsatility.

The Multicenter Study of MagLev Technology in Patients Undergoing Mechanical Circulatory Support Therapy with HeartMate 3 (MOMENTUM 3) trial 2-year data demonstrated an absence of confirmed pump thrombosis requiring pump exchange and marked reduction in stroke rates. On the backdrop of conventional anticoagulation protocols used in the study, observed bleeding complication rates in HM 3 were reduced, yet there is a need for further improvement as the overall intensity of conventional anti-thrombotic therapy represents a major contributor to non-surgical bleeding-related outcomes.

The HM3 LVAS Instructions for Use (IFU) recommend maintaining patients on Warfarin and Aspirin for long-term anticoagulation therapy. Recent results of The Minimal AnticoaGulation EvaluatioN To aUgment heMocompatibility (MAGENTUM 1) pilot study has demonstrated substantially lower-intensity anticoagulation (INR range 1.5 - 1.9) is achievable and supports the safety of lower targets with select patients implanted with the HeartMate 3 beyond 1 year with no thromboembolic complications or pump thrombosis. The observed outcomes were similar to those with the higher intensity anticoagulation targets and further support a signal of enhanced intrinsic thromboresistance of the HM3.

Direct oral anticoagulants (DOACs) are a class of drugs which directly exert therapeutic effect on specific coagulation factors. Broadly, they can be categorized as direct thrombin inhibitors (dabigatran) and factor Xa inhibitors (apixaban, rivaroxaban, and edoxaban) or FXai. Warfarin, which inhibits vitamin K dependent synthesis of coagulation factors in a manner that prevents activation of these factors, has wide inter-individual variation in metabolism and a narrow therapeutic window, as well as both food-drug and drug-drug interactions; the result is that patients taking warfarin require frequent monitoring of the anticoagulant effect to maintain safety and efficacy. The DOAC directly enter the blood to bind to the activated coagulation factor target; they have predictable pharmacokinetics, little interindividual variation in metabolism, few drug-drug interactions, and no interactions with foods. The large phase 3 RCT in both AF and VTE established both efficacy and safety-without the need for monitoring. The FXai may provide better anticoagulation than the oral direct thrombin inhibitor due to their action earlier in the coagulation cascade prior to the generation of thrombin which may ameliorate the likelihood of initiation of the feedback loop resulting in >1000-fold increase in thrombin production. Of the studied FXai , apixaban has the lowest major bleeding complication rate and has not been shown to increase GI-bleeding. It also has the least dependence on renal clearance.

Consequently, with the documented enhanced hemocompatibility of the HeartMate 3 and the potential for reduced major bleeding with apixaban in indicated patient populations, the investigators provide the rationale that patients with the HM3 are in clinical equipoise to be randomized in a feasibility study of a new antithrombotic strategy testing apixaban with or without aspirin compared to the current standard of care warfarin and aspirin in a rigorously structured study to evaluate safety in stable patients with the HM3 device.

Apixaban Safety and Efficacy Data Apixaban is a DOAC that directly inhibits Factor Xa (FXai) in the coagulation cascade. Its therapeutic effect is more consistent and predictable due to its mechanism of action, and it is not subject to the disadvantages inherent to Vitamin K antagonist (VKA) anticoagulants.

The rationale for Apixaban use with the HeartMate 3 There have been no studies to date that have systematically evaluated the feasibility of using apixaban alone or combined with low dose aspirin in HM3 patients. All the primary phase 3 clinical trials assessing DOACs have focused on patients with non-valvular atrial fibrillation or venous thromboembolism with or without cancer. Within the literature, there are sparse reports of apixaban use with LVAD patients due to recurrent bleeding or non-compliance with warfarin. These small sample size studies reported encouraging low rates of thromboembolic events. In all but one instance, aspirin was withheld due to the history of bleeding events. Patients in these studies either had the HeartMate II or HeartWare HVAD.

Reduction in bleeding and thromboembolic events with HeartMate 3 compared to the HeartMate II was demonstrated by the MOMENTUM 3 IDE Trial. Yet, bleeding complications remain a burdensome limitation while on support and represent a significant cause of rehospitalizations and morbidity. Independently, both a reduction in major bleeding events and stable anticoagulation intensity constitute a compelling potential benefit of a modified antithrombotic strategy with a direct oral anticoagulant. However, these apixaban associated benefits remain to be validated in advanced heart failure population supported with the HeartMate 3 LVAS. Therefore, the objective of this study is to assess safety and feasibility of apixaban use in HM3 supported patients.

DATA COLLECTION & FOLLOW-UP ASSESSMENTS The patient will be assessed at baseline. Lactate dehydrogenase (LDH) will be assessed once a week for 4 weeks, then once every 2 weeks for the next month and monthly thereafter; TTE ECHO follow-up will be performed at baseline, at 1 month and at 3 months, followed until study completion per site standard of care.

Study duration Patients enrolled will be followed-up for 90 days post-transition to a designated antithrombotic regimen based on randomization. Provided the individual patients clinical course is uneventful regarding the primary endpoint, the patient's follow-up within the antithrombotic study protocol will be extended to the next pre-specified time point for analysis at 180 days. After the 180 days timepoint is reached, the patients will be given a chance to prolong the study until 1 year ( study extension, approved by Institutional Ethics Commitee on 10-12-2022, approval number: 27261/22; A-21-23). All apixaban subsets will be treated according to their original study arm, the patients from the Vitamin K antagonist and aspirin group will be randomized in a 1:1 manner to apixaban with or without aspirin.

If the individual uneventful primary safety endpoint is established, the patient follow-up will be prolonged with next pre-specified time point for analysis at 1 year. If the second safety endpoint is reached, the patients could be followed for the duration of support with the HeartMate 3. (second study extension, approved by Institutional Ethics Commitee on 05-10-2023, approval number:16047/21; A-21-23).

Advanced Pump Thrombosis Monitoring Protocol

* Monitor LDH at baseline and after initiation of determined antithrombotic therapy based on randomization algorithm once a week during first 4 weeks, then once every 2 weeks for the next month and monthly after that
* If LDH rises more than 1.2x baseline:

  * repeat LDH within the next 1-3 business days
  * monitor plasma free hemoglobin (pf-Hb) and haptoglobin if available; and total bilirubin
  * complete evaluation with the team to rule out other reasons for LDH rise
  * echocardiogram to evaluate for aortic insufficiency
  * prompt study team to review within 48 hours
  * retrospective data log files analysis (particularly rotor noise and rotor displacement trends) followed by prospective analysis 2 weeks post event

ELIGIBILITY:
Inclusion Criteria:

* The patient has been implanted with HeartMate 3 LVAS
* The patient is, at a minimum, 3 months post HeartMate 3 implant
* The patient is stable, ambulatory, and has been discharged home
* The patient provides written informed consent before any clinical investigation related procedure

Exclusion Criteria:

* Non-compliance with anticoagulation and antiplatelet medication, in the opinion of the investigator
* Weight ≤ 60 kgs. or age ≥ 80 years
* Poor kidney function with serum creatinine ≥ 221umol/L or creatinine clearance < 0.042 mL/s, or the need for chronic renal replacement therapy
* Total bilirubin > 43 umol/L, shock liver, or biopsy-proven liver cirrhosis
* Absence of an informed consent
* Presence of any mechanical prosthetic valve or any ancillary circulatory assist device system (other than the HM3)
* Recent history of cardioembolic stroke
* Hemodynamically significant carotid arteries stenosis (documented by imaging investigation not older than 12 months)
* Need for antiplatelet therapy for reasons other than LVAD therapy
* Major HRAE event after HeartMate 3 index hospitalization discharge
* Known history of hyper- or hypo- coagulable disorder
* Anti-phospholipid syndrome positive patients with documented history of thrombotic/thromboembolic events
* Known hypersensitivity or allergy to apixaban or aspirin
* The patient is involved in another interventional study or any study that could potentially affect the functioning of the HM3 LVAD or the therapeutic effect of any of the study anticoagulants (warfarin, apixaban or aspirin), or could potentially confound the study results
* The patient is currently pregnant, breastfeeding, or intending to get pregnant during the study
* Presence of other anatomic or comorbid conditions, or other medical, social, non-compliance or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements or impact the scientific soundness of the clinical investigation results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Netuka, MD, PhD, Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

RESULTS

PARTICIPANT FLOW:
Groups:
- Apixaban Alone Group: This study group contained 16 patients that were given only apixaban 5mg twice a day.
- Apixaban + Aspirin Group: This group contained 15 patients that were given apixaban 5 mg twice a day + aspirin 100mg a day.
- Warfarin + Aspirin Group: This study group contained 14 patients that were treated following standard anticoagulation protocol (Warfarin INR 2-3 + aspirin 100mg/day).
Period: 3 Months
Arm/Group | Apixaban Alone Group | Apixaban + Aspirin Group | Warfarin + Aspirin Group
Started | 16 | 15 | 14
Completed | 15 | 13 | 13
Not Completed | 1 | 2 | 1
Period: 6 Months
Arm/Group | Apixaban Alone Group | Apixaban + Aspirin Group | Warfarin + Aspirin Group
Started | 15 | 13 | 13
Completed | 13 | 9 | 12
Not Completed | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Patients randomized to apixaban group were then randomized in 1:1 ratio in two subgroups - apixaban alone (16 patients) and apixaban + aspirin (15 patients).
Groups:
- Apixaban + Aspirin Group: This study group contained 15 patients that were given apixaban 5mg twice a day + aspirin 100mg a day.
- Total: Total of all reporting groups
Arm/Group | Apixaban Alone Group | Apixaban + Aspirin Group | Warfarin + Aspirin Group | Total
Number analyzed (Participants) | 16 | 15 | 14 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 6 | 22
  >=65 years | 7 | 8 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (11.1) | 59.7 (16.3) | 64.6 (10.8) | 61.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5
  Male | 15 | 13 | 12 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 16 | 15 | 14 | 45
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Czechia | 16 | 15 | 14 | 45

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Hemocompatibility Related Adverse Events During Apixaban Use With the HeartMate 3 LVAS
Description: Evaluation survival free of major hemocompatibility related adverse events (HRAEs). Major HRAEs include:
  * Stroke (ischemic/hemorrhagic)
  * Pump thrombosis
  * Severe bleeding (see Appendix II)
  * Peripheral arterial thromboembolic events Comparison of HRAEs in apixaban and control group per protocol. Separate analysis in patients randomized to receive aspirin and no-aspirin within the apixaban group as specified in protocol.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Apixaban Alone Group: This study group included 16 patients that were given apixaban 5mg twice a day.
- Apixaban + Aspirin Group: This study group included 15 patients that were given apixaban 5 mg twice a day and aspirin 100mg per day.
- Warfarin + Aspirin Group: This study group contained 14 patients treated following standard anticoagulation protocol (Warfarin INR 2-3 + aspirin 100mg/day).
Arm/Group | Apixaban Alone Group | Apixaban + Aspirin Group | Warfarin + Aspirin Group
Number analyzed (Participants) | 16 | 15 | 14
Participants | 0 | 1 | 2

2. Secondary Outcome: Evaluation of Adverse Events Defined by INTERMACS Definitions
Description: The events evaluated are as follows:
  * Stroke (ischemic/hemorrhagic)
  * Pump thrombosis
  * Major bleeding
  * GI Bleeding
  * Peripheral arterial thromboembolic events
  * Transient ischemic attack
  * Hemolysis
  * Venous thromboembolism
  * Myocardial infarction
  * Right heart failure
  * Cardiac arrhythmias
  * Liver and kidney dysfunction
  * Death due to any cause
Time Frame: Through study completion, an average of 1 year.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Apixaban Alone Group: This study group contained 16 patients that were given apixaban 5mg twice a day.
- Apixaban + Aspirin Group: This study group contained 15 patients that were given apixaban 5mg twice a day and aspirin 100mg per day.
Arm/Group | Apixaban Alone Group | Apixaban + Aspirin Group | Warfarin + Aspirin Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 4/16 | 4/15 | 8/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban Alone Group (N=16) | Apixaban + Aspirin Group (N=15) | Warfarin + Aspirin Group (N=14)
GI bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Driveline infection (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hypovolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Right heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Hip luxation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Positive blood cultures (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — One episode of epistaxis requiring treatment

LIMITATIONS AND CAVEATS:
Our study is limited by its single-center design, small numbers and short follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Version 1.0 (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT04974684/Prot_000.pdf
  • Study Protocol: Version 2.0 (2022-09-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT04974684/Prot_001.pdf
  • Study Protocol: Version 3.0 (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT04974684/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT04974684/SAP_004.pdf